CLINICAL TRIAL: NCT02062866
Title: Intradermal Purse-String Closure Vs Second Intention Healing
Brief Title: Evaluation of Purse-String Closure Vs Second Intention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 407301
Record Dates: First submitted 2013-11-01; First posted 2014-02-14 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Wound Closure Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purse-String (Active Comparator): Surgical wounds are healed via suturing.
  Interventions: Procedure: Purse-String; Procedure: Second Intent
- Second Intent (Active Comparator): Surgical wounds are allowed to heal without sutures.
  Interventions: Procedure: Purse-String; Procedure: Second Intent

INTERVENTIONS:
Procedure: Purse-String — The wound will be closed using one, long, continuous suture which will enter and exit run through the skin along the inner edge of the wound. The start and stopping point will be adjacent to one another. The suture will then be pulled" on either side to essentially cinch down the wound, decreasing the size of the wound.
Procedure: Second Intent — The wound will not be sutured, and allowed to heal on its own.

SUMMARY:
To compare healing time, scar size, aesthetic outcome, and complication rates following second intention healing or purse string closure of surgical wounds on the trunk or extremities. This study, will allow surgeons to make informed decisions on whether purse string closure is superior to that of second intention healing and thus worth considering or inferior and not worth performing.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to give informed consent themselves
* Willing to return for follow-up visits
* Post-operative defects greater than 8 mm (in greatest diameter or length of circular or oval geometric shape) on the trunk and extremities (including the shin, hands, and feet)

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Unwilling to return for follow-up
* Pregnant women
* Wounds less than 8 mm in length
* Wounds on the head, neck or digits
* Patients in which primary linear closure is recommended

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Assessment of Scar on the Patient and Observer Scar Assessment Scale | 3 months
  After surgical procedure, subjects will be randomized into one of two wound healing groups: by second intention (no sutures) or by purse-string closure (with sutures). After 3 months, subjects will return to clinic for evaluation of the pain scale and cosmesis of both types of healing techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Dept. of Dermatology, Sacramento, California, United States

REFERENCES:
- [Derived] Joo J, Custis T, Armstrong AW, King TH, Omlin K, Kappel ST, Eisen DB. Purse-string suture vs second intention healing: results of a randomized, blind clinical trial. JAMA Dermatol. 2015 Mar;151(3):265-70. doi: 10.1001/jamadermatol.2014.2313. PMID 25372450
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical